CLINICAL TRIAL: NCT02840422
Title: Assessment of Patients Quality of Life Suffering From Knee Osteoarthritis Treated With Three Intra-articular Injections of ARTHRUM H 2% Over a Period of Six Months
Brief Title: Assessment of Patients Quality of Life Treated With Three ARTHRUM H 2% Joint Injections
Acronym: ART-QUALIVIE
Status: Completed | Type: Observational
Sponsor: LCA Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 140515
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic acid; Knee osteoarthritis; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ARTHRUM H 2% — ARTHRUM H 2%

SUMMARY:
The reduction of functional limits and disablilities induced by knee osteoarthritis as well as improvement of patients quality of life is a public health need registered amongst the priorities established by the French law of August 9th 2004 relative to Public Health policy. However, the response to this need is not limited to treatment with health products.

This clinical trial in real life on ARTHRUM H 2% device aims to analyse patients quality of life treated by intraarticular injections, eventually for several years, by difference of usual clinical trials.

This open, prospective, multicentric study aims to analyse, in patient care, the impact of three intraarticular injections of ARTHRUM H 2% on quality of life over a period of 6 months (D180) in the symptomatic treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Parameters used to determine treatment outcomes include: "Short-Form 12 Health Survey" (SF-12), Pain score of the Western Ontario McMaster Universities Osteoarthritis Index (WOMAC A)

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged over 40;
* Suffering from symptomatic knee osteoarthritis radiologically confirmed less than 12 months ago and stage I, II or III according to KELLGREN (knee in extension) and with minimal pain on walking (WOMAC A1) of two points on the LIKERT scale
* Patient able to understand the trial procedure and give his/her consent to take part, in writing;
* Patient geographically stable during the trial;
* Patient affiliated to the French social security regime or benefiting from such a French regime.

Exclusion Criteria:

* Inflammatory arthritis;
* Progressive infectious condition of the knee being studied;
* Previous treatment with viscosupplementation for at least one year;
* Injection of corticoids into the knee studied for less than two months;
* Known hypersensivity to hyaluronic acid or substances with similar activity;
* Pregnant or breast-feeding women;
* Patient under guardianship or tutorship or under juridicial protection;
* Patient currently taking part in another clinical research study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or Women aged aver 40 ans suffering fromm knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
To measure the physical component summary (PCS) improvement, on patient quality of life suffering from knee osteoarthritis after treatment by three intraarticular injections of ARTHRUM H 2% from D0 (inclusion) to D180 (end of trial) | 6 months

SECONDARY OUTCOMES:
To study quality of life variation, "Short-Form 12 Health Survey" (SF-12) on physical component summary (PCS) | 6 months
  * From D0 to D90
  * From D90 to D180
To study quality of life variation, "Short-Form 12 Health Survey" (SF-12) on mental component summary (MCS) | 6 months
  * From D0 to D90
  * From D0 to D180
  * From D90 to D180
To study pain variation of score A from Western Ontario McMaster Universities Osteoarthritis (WOMAC A) | 6 months
  * From D0 to D90
  * From D0 to D180
  * From D90 to D180

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTIAN PASCARETTI, MD, Study Director — Le Ronceray Rhumatologie; Paolo INSALACO, MD, Study Director — Le Ronceray Rhumatologie; ANTOINE LESORT, MD, Study Chair — Hopital Prive des Peupliers

IPD SHARING:
Plan to Share IPD: No